CLINICAL TRIAL: NCT03361085
Title: Modular Prevention Bundle for Non-ventilator-associated Hospital-acquired Pneumonia (nvHAP)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-Epidemic with changes in patient mix, restructuring of wards/departments, new standard-precautions
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: UHZ nvHAP Bundle
Record Dates: First submitted 2017-10-30; First posted 2017-12-04 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Hospital-acquired Pneumonia; Healthcare Associated Infection; Infection Prevention
Keywords: non-ventilator-associated hospital acquired pneumonia; Hospital-acquired Pneumonia; Healthcare Associated Infection; Adherence; infection prevention; implementation
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Cross Infection

STUDY DESIGN:
Intervention Model Description: quasi experimental intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): nvHAP-Prevention Bundle
  Interventions: Procedure: nvHAP Prevention Bundle

INTERVENTIONS:
Procedure: nvHAP Prevention Bundle — oral care, (early) mobilization, diagnosis and treatment of dysphagia, respiratory physiotherapy, stop Proton pump Inhibitors (PPI) if reasonable

SUMMARY:
Background: Hospital acquired pneumonia (HAP) is divided in two distinct groups, ventilator-associated pneumonia (VAP) and non-ventilator-associated HAP (nvHAP). Although nvHAP occurs more frequently than VAP and results in similar mortality and costs, prevention guidelines and prevention focus almost exclusively on VAP. Scientific evidence about nvHAP prevention is scarce. Therefore, we designed a mixed-methods study to investigate the effectiveness of a newly developed nvHAP prevention bundle and factors that influence its implementation.

Methods: This single-centre project at the 950-bed University Hospital Zurich (UHZ) will engage the wards of nine departments with substantial nvHAP rates. The nvHAP bundle consists of five primary prevention measures: 1) oral care, 2) identification and treatment of patients with dysphagia, 3) mobilization, 4) stopping unnecessary proton pump inhibitors, and, 5) respiratory therapy. Implementation includes the engagement of department-level implementation teams, who sustain the 'core' intervention components of education, training, and environmental restructuring and adapt the implementation strategy to local needs. The effects of the implementation will be analysed by a mixed-method approach. As primary outcome, nvHAP incidence rates will be analysed by Poisson regression models to compare incidence rates before, during, and after the implementation phases (on the hospital and department level). In addition, the association between process indicators and nvHAP incidence rates will be analysed using longitudinal Poisson regression models. A longitudinal, qualitative study and formative evaluation based on interviews and focus groups identifies supporting or hindering factors for implementation success in participating departments dynamically over time. This accumulating implementation experience will be constantly fed back to the implementation teams and thus, represents an active implementation element.

Discussion: This comprehensive mixed-methods study is designed to accomplish both, measure the effectiveness of a new prevention bundle against nvHAP and provide insights into how and why it worked or failed. The results of this study may contribute substantially to patient safety in the area of a rediscovered healthcare-associated infection - nvHAP.

DETAILED DESCRIPTION:
Methods

Aim:

With this mixed-methods study, we aim to investigate the impact of the implementation of a newly designed nvHAP prevention bundle on the nvHAP incidence rate among inpatients in our tertiary care hospital. We will quantify the adherence to the individual bundle elements and qualitatively identify the factors that influence successful implementation.

Objectives:

1. To determine the nvHAP bundle effectiveness on the nvHAP incidence rate
2. To determine the adherence the nvHAP bundle and each of the bundle elements
3. To relate adherence to nvHAP bundle elements with nvHAP incidence rate
4. To qualitatively monitor changes and identify trends in implementation outcomes throughout the study periods
5. To identify which factors in the implementation setting are associated with the actual degree of local implementation of the nvHAP bundle

Study setting:

The study is conducted at the University Hospital Zurich (UHZ), Switzerland, a 950-bed tertiary-care teaching hospital covering all medical specialties except paediatrics and orthopaedics.

Study population:

The study population consists of all patients hospitalized in nine predefined medical and surgical departments and their corresponding wards chosen based on the following criteria; 1) nvHAP rate above the 50th percentile according to UHZ nvHAP data from the year 2017; 2) high absolute number of patients with nvHAP according to UHZ nvHAP data from the year 2017; 3) organizational structure, e.g. departments sharing same nursing or medical personnel; 4) representing both medical and surgical specialties.

Intervention:

The nvHAP bundle: The University Hospital Zurich nvHAP bundle was designed by an interprofessional and interdisciplinary group of experts. Elements were chosen based on the evidence, although scarce, of their effectiveness and based on their anticipated feasibility and implementability. The bundle consists of five prevention measures (details see Annex nvHAP Bundle).

1. Oral care, i.e. mechanical and pharmacological oral care
2. Identification and treatment of patients with dysphagia, i.e. by applying a 'modified swallowing assessment' (MSA) adapted from the 'Standardized Swallowing Assessment' by Perry et al. (15) (Annex 'MSA Perry')
3. Mobilization, i.e. mobilization at least twice daily
4. Stopping unnecessary PPI and antacids
5. Respiratory therapy As not all bundle elements apply to all patients, the patients will first be assessed for indication of the respective prevention measure after admission, clinical deterioration, and major surgery during hospital stay. The execution of the bundle element has to be documented in the electronic medical record (EMR).

Implementation strategy and formative evaluation: Our implementation strategy is designed to increase ownership and local adoption in each department by engaging local implementation teams, who establish department-specific actions based on local needs. This strategy is also intended to facilitate adaptability, i.e. the degree to which the intervention can be adapted to meet local needs (16, 17). Based on an initial behavioural analysis informed by sensitizing frameworks (see below, "Implementation Frameworks") (16, 18, 19), we identified the following as promising intervention functions to increase adherence to the nvHAP bundle: increasing knowledge and understanding about the nvHAP bundle elements through education; imparting skills through technical training; and changing the physical context to increase awareness and support performance of nvHAP measures through environmental restructuring. Whereas these intervention functions to increase adherence to the nvHAP bundle elements make up the foreseeable core intervention components, each department is encouraged to adapt the delivery of these components and to employ additional promotional components according to local context, making up the 'soft periphery' of the intervention.

Local implementation teams, composed of one nurse, one physician and one physiotherapist, will be established in each department. During recurrent "action plan" meetings, the local implementation team from each department, with support from the nvHAP study team, will be responsible for assessing the current implementation status with respect to each bundle element and establishing an "action plan" with a list of planned actions aimed to increase adherence to bundle elements according to local needs. Local implementation teams will be responsible for implementing the nvHAP bundle in their respective departments. Established "action plans" will be revisited to assess progress and refine necessary actions, as described below.

The nvHAP study team, based in the infection prevention department, will form a central coordinating team to provide local teams with support, example training materials, and feedback on process and outcome data. Additionally, we will employ a formative approach, during which we aim to continuously identify influences on implementation efforts (e.g. barriers and facilitators) and feed these insights back to local implementation teams to optimize the potential for implementation success (20). This formative evaluation will occur in stages throughout the project, as described by Stetler and colleagues (20) and presented in Table 1. The formative evaluation will rely primarily on "action plan" meetings as an opportunity to feed information back to local implementation teams regarding identified barriers and facilitators to implementation and to refine implementation action plans accordingly.

Study design:

This mixed methods study collects and analyses quantitative and qualitative data collected during the three study periods (baseline, implementation, and intervention period).

Study periods:

Baseline period will start at the same time for all departments and will be of different length (minimum 12 months) as implementation of nvHAP prevention measures will occur at the department level and the start of implementation activities is chosen by every department, primarily relying on availability of resources.

We define three study periods on the department level, 1) department baseline period, before implementation of nvHAP bundle in the specific department; 2) department implementation period, a two month time frame starting with the beginning of implementation activities in the respective department; 3) department intervention period following the department implementation period.

On the hospital level the three periods are defined as follows: 1) hospital baseline period, before starting implementation in the first department; 2) hospital implementation period, from the beginning of the implementation period of the first department until end of implementation period of the last included department; 3) hospital intervention period following the hospital implementation period.

Implementation framework:

Our study is theoretically informed by the Consolidated Framework for Implementation Research (CFIR) (16) and the Theoretical Domains Framework (TDF). Both the CFIR and the TDF integrate findings from theoretical literature into synthesized frameworks consisting of constructs that may mediate behaviour change. Whereas the TDF domains represent a set of constructs related to individual behaviour change, the CFIR domains include constructs relating to broader organizational behaviour change. For the current inquiry, we find the use of both frameworks useful to capture influencers of behaviour at the individual level, as well as the department, the overall hospital, and the wider environmental context. The CFIR and the TDF will inform the intervention implementation strategy, as previously described, and guide the qualitative data collection (semi-structured interview guides) and analyses (use of TDF as deductive coding framework). In particular, use of these sensitising frameworks throughout our study will facilitate the timely identification of barriers and facilitators and will also provide insights as to which additional intervention components are most likely to be successful in addressing the identified barriers.

Data collection:

Data sources: In the study hospital, all patient data are charted electronically via an EMR system. Selected data are stored in a clinical data warehouse.

NvHAP surveillance We apply the European Centre for Disease Prevention and Control (ECDC) definition criteria for pneumonia that are used in the ECDC point prevalence studies (10) (Annex 'ECDC Definition nvHAP') and a validated semi-automated surveillance system for nvHAP is used (22). Place of nvHAP acquisition is defined as department, ward and room to which the patient was affiliated 48h before first symptoms of nvHAP, unless shorter incubation period was evident from patient history.

Process indicators:

Process indicators portraying adherence to the nvHAP bundle elements will be monitored in two ways. First, for all five prevention measures, at least one surrogate parameter for adherence is continuously extracted from the EMR of the total patient population (continuous process indicators; see Annex 'Process indicators'). This parameter, e.g. toothbrushing provided by nurses, will be expressed per department, and month, and either hospital days or admissions. Second, we will monitor process indicators on a sample basis with individual assessment of a subset of patients at four different time points per department (intermittent process indicators; see Annex 'Process indicators'). The latter allows a more detailed description of adherence, including non-documented prevention measures (e.g. oral care executed by patient) and takes into consideration the individual need of patients for the specific prevention measure (e.g. respiratory therapy is indicated only in a subset of patients). From the intermittent process indicators the 'nvHAP adherence score' will assess patient based adherence per department and time point. The score is based on samples of 50 patients, the 'nvHAP adherence indicator' takes the value 1 in the case the specific prevention measure was completed in the specific patient, 0 if that was not the case, and "empty" in the case of missing values. The 'nvHAP adherence score' is calculated by summing up the five proportions of patients with completed specific prevention measures (i.e. 'nvHAP adherence indicator'=1) dividing it by factor five (Annex 'nvHAP adherence score').

Qualitative data collection:

Longitudinal qualitative data will be collected throughout the project as portrayed in Figure 2, including action plan interviews with local implementation teams, drop-in interviews with frontline staff, and focus group interviews, as described in Table 2. These three data collection activities will allow for rigorous triangulation of findings among data sources and will all inform the ongoing formative evaluation (see Table 1).

ELIGIBILITY:
The study population consists of all patients hospitalized in nine predefined medical and surgical departments and their corresponding wards chosen based on the following criteria

* nvHAP rate above the 50th percentile according to UHZ nvHAP data from the year 2017
* high absolute number of patients with nvHAP according to UHZ nvHAP data from the year 2017
* organizational structure, e.g. departments sharing same nursing or medical personnel
* representing both medical and surgical specialties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45000 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
nvHAP Incidence rate | up to 3 months post-discharge
  non Ventilator-associated Hospital acquired Pneumonia according to ECDC definitions

SECONDARY OUTCOMES:
Percentage of patients who passed away during hospitalization (in-hospital mortality) | up to 3 months post-discharge
  death during hospitalisation
length of stay | up to 3 months post-discharge
  Duration of hospitalisation

OTHER OUTCOMES:
Percentage of patients in whom the respective prevention measure was correctly applied (prevention measures are: oral care, mobilisation, dysphagia screening, stopping proton pump inhibitors, respiratory therapy) | at four timepoints (baseline, 2-3 months 4-6 months and 10-12 months after start implentation, 10
  Aderence to the five prevention measures: oral care, Identification and treatment of patients with dysphagia, mobilization, Stop proton pump inhibitors if not indicated, respiratory physiotherapy
Adherence score per department and timepoint | at four timepoints (baseline, 2-3 months 4-6 months and 10-12 months after start implentation, 10
  The 'nvHAP adherence score' is calculated by summing up the five proportions of executed prevention measures (i.e. nvHAP adherence indicator = 1) and dividing it by factor five. In the above example it would be (32/45 + 20/50 + 48/50 + 42/50 + 24/32)/5 = 0.732.
Implementation success evaluated by semi-structured interview and focus group interview | at three timepoints ( 2-3 months 4-6 months and 10-12 months after start implentation, 10
  We will use a qualitative definition of implementation success composed of the following four implementation outcomes: acceptability, appropriateness, protocol fidelity, and sustainability

CONTACTS AND LOCATIONS:
Overall Officials: Aline Wolfensberger, MD, Principal Investigator — University of Zurich; Lauren Clack, PhD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Dept. of Infectious Diseases and Hospital Epidemiology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wolfensberger A, Clack L, von Felten S, Faes Hesse M, Saleschus D, Meier MT, Kusejko K, Kouyos R, Held L, Sax H. Prevention of non-ventilator-associated hospital-acquired pneumonia in Switzerland: a type 2 hybrid effectiveness-implementation trial. Lancet Infect Dis. 2023 Jul;23(7):836-846. doi: 10.1016/S1473-3099(22)00812-X. Epub 2023 Mar 6. PMID 36893785
- [Derived] Wolfensberger A, Clack L, von Felten S, Kusejko K, Faes Hesse M, Jakob W, Saleschus D, Meier MT, Kouyos R, Held L, Sax H. Implementation and evaluation of a care bundle for prevention of non-ventilator-associated hospital-acquired pneumonia (nvHAP) - a mixed-methods study protocol for a hybrid type 2 effectiveness-implementation trial. BMC Infect Dis. 2020 Aug 17;20(1):603. doi: 10.1186/s12879-020-05271-5. PMID 32807090